CLINICAL TRIAL: NCT06839014
Title: Exercise Therapy in Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Our Lady of the Lake Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#8333_Kansara Exer Therapy
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma HNSCC
Keywords: Exercise Therapy; TENS Unit Therapy; Exercise and Cancer; Exercise and Immune Response
MeSH Terms: conditions — Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cancer Treatment Only (No Intervention): Subjects will undergo their prescribed cancer treatment therapy (radiation/chemo/adjuvant)
- Cancer Treatment + Exercise TENS therapy (Experimental): Subjects will undergo prescribed cancer therapy (chemo/radiation/adjuvant) with the addition of an at-home analog TENS unit exercise therapy regimen
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Perform 30 minutes of TENS unit exercise muscle stimulation each day for 3 days a week for the duration of cancer treatment.
  Arms: Cancer Treatment + Exercise TENS therapy

SUMMARY:
The goals of this clinical trial are to learn 1. Determine the feasibility of a home-based exercise analog therapy using Transcutaneous Electrical Nerve Stimulation (TENS), 2. Determine the effects of exercise analog therapy on muscle mass, strength, and clinical outcomes, and 3. Determine the effects of exercise analog therapy on immune phenotype and inflammation response in patients undergoing radiation for head and neck squamous cell carcinoma (HNSCC).

The main question it aims to answer are:

Does an exercise regimen using an analog TENS unit during the course of cancer treatment for those with HNSCC improve muscle mass, strength, clinical outcomes and immune response compared to those that do not perform the exercise regimen during their cancer treatment?

Researchers will compare outcomes of patients undergoing cancer treatment + TENS unit exercise to those being treated for their cancer with no exercise TENS unit.

In the exercise arm, subjects will use the TENS unit for 30 minutes of exercise a day, 3 times a week for the extent of their cancer treatments.

Weekly check-ins by phone or less frequently at scheduled in person visits.

Participants will keep a log of their exercise sessions to make sure that the exercise occurs 3 times a week for 30 minutes each and note any reasons why a session may have been missed or time shortened.

Both arms will have a blood draw at the beginning of their cancer treatment and approximately 4 weeks after the last cancer treatment (~40mL). These samples will be tested for molecules that signal a higher or lower immune response with the addition of the exercise in one group compared to the cancer therapy only group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older)
* Diagnosed with head and neck squamous cell carcinoma
* HPV negative
* Undergoing treatment at OLOL H&N Center

Exclusion Criteria:

* Any subject less than 18 years of age.
* Subjects who have HPV positive HNSCC
* Subjects who have a pacemaker or electronic implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Patients that complete TENS unit exercise as recommended | beginning of cancer treatment to 4 weeks after cancer treatment concludes
  The documentation of successful completion of exercise with the recommended use guidelines (30min, 3 times a week for duration of cancer therapy) will determine if using this type of low maintenance analog exercise muscle stimulation is practical for use in this patient population.

SECONDARY OUTCOMES:
Body Mass Index (BMI)=Weight (kg)/Height (m)^2 | Once at beginning of cancer treatment and once 4 weeks post-cancer treatment
  Body Mass Index using Height (m) vs Weight (kg) to calculate the BMI once pre cancer treatment and once post cancer treatment/intervention. BMI=Weight (kg)/Height (m)^2. This will identify what the effect of this analog exercise may have on the subject's BMI.
Percent Fat/Water/Muscle Content of Body | Once prior to cancer treatment and once 4 weeks post treatment
  The Fat/Water/Muscle content ratio will be measured in both the control group and the exercise group prior to beginning cancer treatment with our without exercise and then 4 weeks post-treatment using Bioelectrical Impedance Analysis (a scale that a person stands on that measures body content ratios (%) of these three macromolecules). This measurement will also identify the effect of using the TENS unit analog exercise regimen on a subject's overall body composition.
Levels/Amount of Immunophenotypic Molecules from Blood Diagnostics (pg/mL) | Beginning of cancer treatment to 4 weeks post-cancer treatment
  Immune response markers identified in the blood samples taken prior to cancer treatment and post treatment (exercise therapy occurring throughout this timeframe) will determine if the inclusion of this TENS unit exercise increases or decreases an immune response. The molecules identified will be measured in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lebeouf Leboeuf, DNP, Study Director — Our Lady of the Lake Hospital

IPD SHARING:
Plan to Share IPD: No